CLINICAL TRIAL: NCT05538936
Title: The Effect of Spa and Massage on Babies on Colic Symptoms: A Randomised Controlled Trial
Brief Title: The Effect of Spa and Massage on Babies on Colic Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Rıdvan Akdogan, Research Assistant (PhD Candidate), Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Istanbul University-Cerrahpaşa
Record Dates: First submitted 2022-09-01; First posted 2022-09-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Infantile Colic; Infantile Spasm
Keywords: İnfantile Colic; Baby SPA; hydrotherapy; massage
MeSH Terms: conditions — Colic; Spasms, Infantile | interventions — Hydrotherapy; Massage; Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design with pretest-posttest experiment and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baby SPA (Experimental): Baby SPA application time: It is done regularly from the first month, at least once a month. The ideal time for application is the first six months. The water in the tub is prepared to be 33°C. The baby, whose clothes are taken off, wearing a waterproof diaper suitable for the tub and a neck ring, is taken into the tub. The application usually takes 10-15 minutes, depending on the baby's reactions to the water for the first time. After the parent and baby get used to the process, the time can be increased to 30 minutes. In this process, the baby's hands, abdomen, and legs are made to recognize the water and the baby's movements are monitored. Care is taken that the baby does not drink the water. After the application period is over, the baby is removed from the tub and dried with a towel. Finally, the baby is massaged for 10-15 minutes and dressed.
  Interventions: Other: Baby SPA
- Massage (Experimental): Massage can be applied to all age periods. Before starting the massage application in babies, some preparations are made. Ambient temperature (24-26 OC) is adjusted, it is regulated so that there is no airflow, dim light, and low noise levels are ensured. 1-2 towels, a soft cushion or massage table, baby oil lotion, clean diapers, and clean clothes are prepared for the massage. There is no standard time interval for the application of massage. It can be done at least one hour after the baby's feeding, at any time of the day when he is not stressed and sleeps. Massage application time is 15-30 minutes depending on the baby's reactions may vary between.
  Interventions: Other: Massage
- Control (No Intervention): It is the control group in which no intervention was applied.

INTERVENTIONS:
Other: Baby SPA — "Salus Per Aquam", "Sanitas Per Aquam", "Salut Per Aqua" or "Solus Per Aqua" (SPA) means health that comes with water. Baby SPA is a physiotherapy method that stimulates the baby's motor movements through water (hydrotherapy) and performs it in an integrated way to balance the body, mind, and emotions. Baby SPA is applied in specially designed bathtubs. The size of the tub is designed in such a way that children can move their hands and feet freely and not be narrow. A neck ring/ring is used to keep the baby on the water surface during SPA treatment.
  Other Names: Hydrotherapy
  Arms: Baby SPA
Other: Massage — The best way to communicate with a baby is to touch it. When babies are born, unlike their other senses, the most developed one is the sense of touch. Because this process begins while in the womb. The baby communicates by touch and begins to recognize his environment. The sense of touch is a priority for the development of all senses. They need to perceive their environment, especially in newborns and infancy periods. Touching the body in a systematic way for a therapeutic purpose is called "Massage". Massage is soft touches to body tissues to relax muscles, accelerate circulation, reduce infantile colic symptoms and pain, regulate sleep, and increase its duration. Baby massage has many benefits such as reducing colic symptoms, increasing weight gain, providing motor development and coordination, strengthening the parent and baby bond, supporting growth and development, and reducing stress.
  Other Names: Therapeutic Touch
  Arms: Massage

SUMMARY:
Although various complementary health approaches have been examined to alleviate colic symptoms, there seems to be a limited number of studies on SPA and massage applications. For this reason, the study was planned to determine the effectiveness of nurses' baby SPA and massage practices in reducing colic symptoms in babies.

DETAILED DESCRIPTION:
Baby SPA is a physiotherapy method that stimulates the baby's motor movements through water (hydrotherapy) and performs body circulation in an integrated way to balance the mind and emotions. Playing with water, the baby's muscles develop, circulation accelerates and the body becomes flexible. It also increases the intestinal motility of the baby. This allows the baby to pass gas more easily. In addition, all parts of the body of the baby floating in the water develop. Because in the water, the hands and legs move freely, giving the whole body the ability to move. Due to the low gravitational effect while swimming in the water, the baby's ability to control their muscles develops, which allows the baby to move more and all of their muscles to work optimally. On the other hand, when the baby is in the water, he feels that he is in an environment similar to the intrauterine environment he is used to.

Infant massage also used to reduce the symptoms of infantile colic, is often called stimulus touch. Baby massage can be defined as a relaxed conversation between parent and baby. Infant massage is also called touch therapy, which refers to a technique that combines the physical benefits of human touch with emotional benefits such as mind bonding. Massage is an application that makes the baby more sensitive, develops a sense of security, enables better communication with eye contact, increases comfort, creates a deep bond between parent and baby, as well as supports the baby's physical, mental and emotional development.

Although various complementary health approaches have been examined to alleviate colic symptoms, there seems to be a limited number of studies on SPA and massage applications. For this reason, the study was planned to determine the effectiveness of nurses' baby SPA and massage practices in reducing colic symptoms in babies.

ELIGIBILITY:
Inclusion Criteria:

* The willingness of the family to participate in the research
* The baby is between 40 days - 4 months
* The baby was born at term
* Birth weight between 2500 - 4500 g
* The baby's diagnosis of infantile colic by the doctor
* The baby has not started any treatment for infantile colic

Exclusion Criteria:

* The presence of any congenital anomaly in the baby
* The baby has a diagnosis of lactose intolerance
* The baby has an acute or chronic illness
* There is a wound on the baby's skin or a condition that prevents massage.
* Having a situation that prevents communication with the mother

Ages: 40 Days to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Data Collection | 6 or 7 months
  The researcher will collect the research data at Van Aquarium Baby SPA and Van İki Nisan Caddesi Private Clinic Center. For the experimental groups, once a week for a total of four applications, the application will end at the end of a month. Introductory Information Form, Infant Colic Scale, and Infant Colic Symptoms Follow-up Form will be applied to the individuals in the experimental and control groups to collect data. Items in the infant colic scale are graded on a Likert-type score from 1 to 6. The rating ranges from 1 (strongly disagree) to 6 (strongly agree). A low mean score from the scale indicates a decrease in colic, while a high mean score indicates an increase in colic. The Baby Colic Symptoms Follow-up Form is a form that measures the duration and frequency of changes in the baby's colic symptoms. If the time and frequency are reduced, it is concluded that the application is effective.

CONTACTS AND LOCATIONS:
Overall Officials: Rıdvan Akdoğan, PhD, Principal Investigator — Yuzuncu Yil University
Locations (1):
- Yuzuncu Yıl University, Van, Turkey, Turkey (Türkiye)

REFERENCES:
- [Derived] Akdogan R, Yildiz S. The effect of SPA and massage applied on babies on colic symptoms: A randomized controlled trial. J Pediatr Nurs. 2025 May-Jun;82:e164-e174. doi: 10.1016/j.pedn.2025.04.008. Epub 2025 Apr 18. PMID 40253272